CLINICAL TRIAL: NCT06348862
Title: Assessment of Stress and Anxiety for Patients Undergoing MRI Using, Holy Quran, Music, and Natural Sounds: A Double Blinded Parallel Randomized Controlled Study
Brief Title: Assessment of Stress and Anxiety for Patients Undergoing MRI Using, Holy Quran, Music, and Natural Sounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Quds University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 323/REC/2023
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-03

CONDITIONS: Anxiety; Stress; MRI Contrast Media Adverse Reaction
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Listening to Quran (Experimental): Listening to Quran during MRI
  Interventions: Behavioral: Listening to either Quran, Music, and or Natural sound
- Listening to Music (Experimental): Listening to Music during MRI
  Interventions: Behavioral: Listening to either Quran, Music, and or Natural sound
- Listening to Natural Sound (Experimental): Listening to Natural Sound during MRI
  Interventions: Behavioral: Listening to either Quran, Music, and or Natural sound
- Listening to nothing (No Intervention): Listening to nothing during MRI

INTERVENTIONS:
Behavioral: Listening to either Quran, Music, and or Natural sound — Patients will be assigned into one of the four groups based on their preferences. These groups are people who will listen to either Quran, Music, Natural sound, and or nothing (control group).
  Arms: Listening to Music; Listening to Natural Sound; Listening to Quran

SUMMARY:
The aim of the current study is to analyze the effect of listening to Quran or music or natural sounds on anxiety and stress level among patients undergoing MRI.

DETAILED DESCRIPTION:
After informed consents will be obtained from patients undergoing Magnetic Resonance Image (MRI). A randomized Controlled Parallel design will be used to assess the effectiveness of listening to Quran, music, and natural sound to reduce anxiety and stress level among patients undergoing MRI in Palestine. A control group will receive the traditional care during MRI without listening to any sound, while the intervention groups will listen to either Quran, music, or natural sounds during the MRI scan. Notice that each patient will choose the preferred method to be in one of the four mentioned groups. This study will include participants with predetermined specific eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Who agreed to participate in this study.
* Both sex.
* Age of 18 years and above.
* Fully conscious and oriented.

Exclusion Criteria:

* Referrals from the intensive care unit.
* Life-threatening situations.
* General ill health,
* Serious psychological disorders.
* Invasive MR imaging procedures (such as biopsies).
* Being under the age of 18, and
* Exams that were particularly scheduled for other investigations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Level of Anxiety among patients who underwent MRI | Ten to 30 minutes according to the duration of MRI
  Level of Anxiety among patients who underwent MRI
Level of Stress | Ten to 30 minutes according to the duration of MRI
  Level of Stress among patients who underwent MRI

SECONDARY OUTCOMES:
Sociodemographic | Ten to 30 minutes according to the duration of MRI
  If Sociodemographic data such as (age, sex, level of education..etc.) will have an effect on the level of anxiety and stress after listening to the one of the three interventions (Quran, music, or natural sound).

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Quds University, East Jerusalem, Jerusalem, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Yes
Demographics such as age, sex, level of education, income, marital status, if work or not, type of work, if chronic disorder is present.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: April 1, 2025